CLINICAL TRIAL: NCT05861180
Title: Neck Joint Position Error Among Taibah Students University; Saudi Arabia; Cross Section Design
Status: Completed | Type: Observational
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, walaa M Ragab, assistant professor, Taibah University
Other Study IDs: taibah
Record Dates: First submitted 2023-04-29; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Proprioception
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal group: no text neck
  Interventions: Device: inclinometer, smart phone goniometer and laser beam
- mild text neck
  Interventions: Device: inclinometer, smart phone goniometer and laser beam
- moderate text neck
  Interventions: Device: inclinometer, smart phone goniometer and laser beam
- severe text neck
  Interventions: Device: inclinometer, smart phone goniometer and laser beam

INTERVENTIONS:
Device: inclinometer, smart phone goniometer and laser beam — devices to objectively assess proprioception of the neck

SUMMARY:
this study was done to answer the following: Is there a difference between students without and with varying degrees of text neck in cervical proprioception defect? Is there a correlation between JPE and severity of text neck among Taibah students University?

ELIGIBILITY:
Inclusion Criteria:

* A convenient sample of 68 female students
* the age was between 18-25 years

Exclusion Criteria:

* Any students with neck pain or previous neck or back surgery or a history of a previous accident were excluded
* Also, we excluded any student with a history of fracture injury of the cervical column, scoliosis, severe thoracic kyphosis, rheumatic disease, torticollis, loss of standing balance, use of hearing aid, and persistent respiratory problems.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All four groups were recruited from the college of medical rehabilitation sciences, Applied Medical Sciences, and Business administration faculty through posters, word of mouth, and by WhatsApp groups.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
neck proprioception error | one day
  we measured joint position error for all students from sitting and standing using laser beam detection error

SECONDARY OUTCOMES:
joint position error | one day
  we measured joint position error of cervical spine by measuring neck motion by phone goniometer and inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: walaa ragab, phd, Principal Investigator — Taibah University
Locations (1):
- Taibah University, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No